CLINICAL TRIAL: NCT04654195
Title: Associations Between Genetic Polymorphisms of Drug Transporter Genes and Toxicity of Doxorubicin and Cyclophosphamide Chemotherapy in Breast Cancer Patients
Brief Title: Study of ABCB1,SLC22A16 Drug Transporter Genes and Doxorubicin and Cyclophosphamide Toxicity in Brest Cancer Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Damanhour University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Other Study IDs: 0000012
Record Dates: First submitted 2020-04-29; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Patients
MeSH Terms: interventions — Amplified Fragment Length Polymorphism Analysis; Polymorphism, Single Nucleotide; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted by extraction kits from whole blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Genetic: polymorphism analysis — DNA will be purified from whole blood samples by commercial DNA isolation kits. Genotyping and genetic polymorphism detection for some metabolic enzymes genes will be performed by real time PCR.
  Other Names: single nucleotide polymorphism
Drug: Doxorubicin-Cyclophosphamide regimen — Treatment with a combination of Doxorubicin and Cyclophosphamide, This regimen comprises 60 mg/m² Doxorubicin and 600 mg/m² Cyclophosphamide administered intravenously on day 1 of each 21-day cycle, and repeated for a total of four cycles.
  Other Names: chemotherapy treatment

SUMMARY:
polymorphisms of drug transporter genes may influence of Doxorubicin-Cyclophosphamide toxicity in breast cancer patients.

the investigators want to

evaluate the association between associations between genetic polymorphisms of ABCB1,SLC22A16 Genes and Toxicity of Doxorubicin and Cyclophosphamide Chemotherapy in Breast Cancer Patients treated by Doxorubicin-Cyclophosphamide regimen therapy

DETAILED DESCRIPTION:
breast cancer is the most common cancer diagnosed in women .Breast cancer can occur in both men and women, but it's far more common in women.

The etiology of breast cancer possesses a multifactorial origin , showing as risk factors reproductive age, early menarche, late menopause, nulli parity, exogenous hormones ,smoking, obesity, diet, alcohol consumption, physical inactivity, and genetic and environmental factors(1).

Chemotherapy combination usually used in treat breast cancer specially cyclophosphamide which is alkylating agent and doxorubicin which is cytotoxic drug.

Doxorubicin entry to the cell is facilitated by the solute importer SLC22A16,the efflux of AC drugs uses several ATP-binding cassette transporters (ABC),( ABCB1, ABCC1, ABCC2, ABCG2)(2),(7).

Most chemotherapeutic agents are not specific against neoplastic cells , also affecting normal cells. Which result in a wide range of adverse reactions in virtually all tissue of body. Unfortunately, chemotherapy-induced toxicities are commonly affecting cancer patients with various intensity, and could be the reason for treatment delays and significantly lowered quality of life. Hematological and gastrointestinal toxicities are common in patients treated with cyclophosphamide and doxorubicin(3).

Extremely high proliferative capacity of hematopoietic system makes it the collateral target for chemotherapeutic agents. Chemotherapy-induced neutropenia are , because of the high susceptibility of neutrophil lineage to cytotoxic effects of cancer treatment. The drug-induced destruction of neutrophil precursors in bone marrow is the main cause of those symptoms. Decrease in neutrophil count is managed by the dose reduction and delays that decrease the dose intensity, where is maintaining the dose is important for favorable response to treatment(3). Another frequent and serious myelotoxic symptom in breast cancer chemotherapy is anemia. This condition may emerge from the disease itself, but the effect of concomitant administration of cytotoxic drugs is also the cause of drop in the hemoglobin level. Anemia has deleterious effect on patients' quality of life as well as on the treatment response. The suspected causes include blood loss, reduced or impaired erythrocytes production and high rate of red blood cells destruction or their reduced survival(4).

Chemotherapy-induced nausea and vomiting (CINV) is a common severe side effect for cancer patients undergoing emetic chemotherapy. The complete pathophysiology of CINV is not known but gastrointestinal (GI) side effects associated with anticancer chemotherapy are traditionally thought to be attributable to mucosal damage.

Nausea is complex in nature and probably depending on more than one etiological factor . Different pathways have been identified for acute and delayed CINV Also, nausea and vomiting can result in anorexia, decreased performance status, metabolic imbalance, wound dehiscence, esophageal tears and nutritional deficiency(5).

In the study we will focuse on the analysis of the relations between the polymorphic variants in some drug transporter genes with known or potential role in the AC-induced toxicity. Single nucleotide polymorphisms will analyzed in genes encoding proteins Involved in AC drug transport

ELIGIBILITY:
Inclusion Criteria:

1. women who has confirmed diagnosis of breast cancer.
2. patient who will be treated with cyclophosphamide and doxorubicin(AC) regimen only .
3. patient take drug regimen for first time.

Exclusion Criteria:

- 1. Patients with metastatic disease and with other previous tumors were excluded from this study 2. Pregnant or nursing female. 3. The patients who were diagnosed with cardiovascular disease or with low left ventricular ejection fraction.

4 .patients who had benign breast cancers, or had no clinical pathological information

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all breast cancer females reciving (Ac regimen) at El-hosien University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
.1-The frequency of the genetic polymorphisms of ABCB1 in breast cancer patien | up to 24 week
  the blood samples will be DNA extracted using DNA extraction kit then single nucleotide polymorphisms of CYP2C19 gene will be detected by real time PCR
The frequency of the genetic polymorphisms of SLC22A16 in breast cancer patients | up to 24 week
  the blood samples will be DNA extracted by DNA extraction kit then single nucleotide polymorphisms of SL22A16 gene will be detected by real time PCR

SECONDARY OUTCOMES:
Correlation between genetic polymorphisms of ABCB1 and toxicities from Doxorubicin-Cyclophosphamide regimen therapy | up to 24 week
  the blood samples will be DNA extracted using DNA extraction kit then single nucleotide polymorphisms of ABCB1 gene will be detected by real time PCR
Correlation between genetic polymorphisms of SLC22A16 and toxicities from Doxorubicin-Cyclophosphamide regimen therapy | up to 24 weeks
  the blood samples will be DNA extracted by DNA extraction kit then single nucleotide polymorphisms of SL22A16 gene will be detected by real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Hoda salem, Ass.prof, Study Director — Faculty of pharmacy Al-Azhar University for Girls; Wael helmy, Ass.prof, Principal Investigator — Faculty of medicine Al-Azhar University for Boys; Amira bisheer, PhD, Principal Investigator — faculty of pharmacy ,Damanhour University; sanaa mohsen, B.pharm, Principal Investigator — faculty of pharmacy,Al-Azhar University
Locations (1):
- Elhussien University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Tecza K, Pamula-Pilat J, Lanuszewska J, Butkiewicz D, Grzybowska E. Pharmacogenetics of toxicity of 5-fluorouracil, doxorubicin and cyclophosphamide chemotherapy in breast cancer patients. Oncotarget. 2018 Jan 10;9(10):9114-9136. doi: 10.18632/oncotarget.24148. eCollection 2018 Feb 6. PMID 29507678
- [Background] Ludovini V, Antognelli C, Rulli A, Foglietta J, Pistola L, Eliana R, Floriani I, Nocentini G, Tofanetti FR, Piattoni S, Minenza E, Talesa VN, Sidoni A, Tonato M, Crino L, Gori S. Influence of chemotherapeutic drug-related gene polymorphisms on toxicity and survival of early breast cancer patients receiving adjuvant chemotherapy. BMC Cancer. 2017 Jul 26;17(1):502. doi: 10.1186/s12885-017-3483-2. PMID 28747156
- [Background] 3-U.S. department of health and human services(2017): Common Terminology Criteria for Adverse Events (CTCAE),National Cancer Institute ,2017,pp(4-6 ) ,pp(24-44).
- [Background] Islam MS, Islam MS, Parvin S, Ahmed MU, Bin Sayeed MS, Uddin MM, Hussain SM, Hasnat A. Effect of GSTP1 and ABCC4 gene polymorphisms on response and toxicity of cyclophosphamide-epirubicin-5-fluorouracil-based chemotherapy in Bangladeshi breast cancer patients. Tumour Biol. 2015 Jul;36(7):5451-7. doi: 10.1007/s13277-015-3211-y. Epub 2015 Feb 13. PMID 25677905